CLINICAL TRIAL: NCT01913899
Title: Short Term Effect of Post Surgical Treatment of Mirror Therapy of Phantom Limb Pain
Acronym: PPSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Deutsche Gesetzliche Unfallversicherung (DGUV) (Unknown)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof. Dr. Christoph Maier, Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4318-12
Record Dates: First submitted 2013-07-30; First posted 2013-08-01 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2012-04

CONDITIONS: Phantom Limb Pain
Keywords: phantom limb pain; mirror therapy; amputees; phantom limb; occupational therapy
MeSH Terms: conditions — Phantom Limb | interventions — Physical Therapy Modalities; Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirror therapy (Experimental): 60 minutes of mirror therapy each day over a period of 14 days starting directly post surgically (24-48 hours after surgery)
  Interventions: Other: Occupational/ physical therapy; Other: Mirror therapy
- Occupational/ physical therapy (Active Comparator): 60 minutes of occupational/ physical therapy each day over a period of 14 days starting 24-48 hours post surgically
  Interventions: Other: Occupational/ physical therapy

INTERVENTIONS:
Other: Occupational/ physical therapy
Other: Mirror therapy — - Intervention group: treatment sessions of 60 minutes with mirror therapy over a period of 14 days starting directly post surgical (24-48 hours)
  Arms: Mirror therapy

SUMMARY:
The aim of the study is the measurement of the short term effect of post surgical mirror therapy concerning pain intensity and frequency of patients with upper or lower amputation in comparison to standard occupational or physical therapy. The hypothesis is that patients in the intervention group (mirror therapy) suffer significantly less from phantom limb pain and pain attacks within a follow-up period of 4-8 weeks.

DETAILED DESCRIPTION:
Aim:

* Measurement of the short term effect of post surgical/ post-operative mirror therapy concerning pain intensity of patients with upper or lower amputation in comparison to standard occupational/ physical therapy
* Hypothesis: patients in the intervention group (mirror therapy) suffer from significant less phantom limb pain and a lower pain frequency within a follow-up period of 4-8 weeks

Methods:

* Design: multicenter, prospective, randomized controlled trial
* Participants: 70, 35 per intervention and con-trol group
* Intervention group: treatment sessions of 60 minutes with mirror therapy over a period of 14 days starting directly post surgical (24-48 hours)
* Control group: receive treatment session of 60 minutes with the same treatment frequency over a period of 14 days
* Measurement tools:

Primary objectives

* pain intensity (11 point NRS, phantom limb in-tensity)
* pain frequency (amount of pain attacks) Secondary objectives
* diary
* daily assessment of mirror and physical thera-py sessions
* analysis:
* in significant differences between the groups a covariance analysis will be performed
* comparison of medians

ELIGIBILITY:
Inclusion Criteria:

* major amputation of lower and upper body
* phantom pain, or pain attacks in combination with a treatment wish
* age of 18 years
* signed informed consent
* linguistic and cognitive comprehension

Exclusion Criteria:

* bilateral amputation
* major neurologic comorbidities (stroke, Parkinson disease)
* morbidities of the contralateral side with functional limitations
* experience with long term standardised mirror therapy
* internal comorbidities (pAVK)
* psychological comorbidities

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Current pain intensity | after 14 treatment sessions
  Current Pain intensity assessed by the Numeric Rating Scale (0-10)

SECONDARY OUTCOMES:
Frequence of pain attacks | after 14 treatment sessions
  Total number of phantom limb pain attacks per day is documented

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, Prof. Dr., Principal Investigator — Ruhr University Bochum; Andreas Schwarzer, Dr. Dr., Principal Investigator — Ruhr University of Bochum
Locations (1):
- Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil GmbH, Bochum, North Rhine-Westphalia, Germany